CLINICAL TRIAL: NCT02416479
Title: SystemCHANGE: An Intervention for Medication Adherence in Transplant Recipients
Brief Title: SystemCHANGE: An Intervention for Medication Change in Adult Kidney Transplant Patients
Acronym: MAGIC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cynthia Russell (Other)
Collaborators: University of Tennessee (Other); University of Missouri-Columbia (Other)
Responsible Party: Sponsor-Investigator, Cynthia Russell, Professor, University of Missouri, Kansas City
Organization: University of Missouri, Kansas City (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0039040
Record Dates: First submitted 2015-04-04; First posted 2015-04-15 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Kidney Disease
Keywords: medication adherence; outcomes; intervention; randomized controlled trial
MeSH Terms: conditions — Kidney Diseases; Medication Adherence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SystemCHANGE (Experimental): SystemCHANGE supports patient-designed, interventionist-guided, small experiments to: 1) assess individual systems (including important others who shape medication taking) and the system's impact on medication taking and propose individual system solutions to improve MA, 2) implement the proposed individual systems' solutions to improve MA, 3) track MA data, and 4) evaluate MA data.
  Interventions: Behavioral: SystemCHANGE
- Patient-education attention-control (Active Comparator): The 6-month Patient education attention-control (AC) intervention includes 6 transplant educational materials, covering healthy post-transplant behavior, developed by the International Transplant Nurses Society. The RA calls Pps at 1, 2, 3, 4, 5 and 6 months to review the brochure information and answer any questions about it.
  Interventions: Behavioral: Patient-education attention control

INTERVENTIONS:
Behavioral: SystemCHANGE — SystemCHANGE self-management supports patient-designed, interventionist-guided, small experiments using Deming's Plan-Do-Check-Act cycle26 to: (1) assess individual systems (including important others who shape medication taking), how they influence medication taking and their proposals for improving medication adherence, (2) implement the proposed individual systems' solutions to improve adherence, (3) track adherence data, and (4) evaluate adherence data.
  Arms: SystemCHANGE
Behavioral: Patient-education attention control — The 6-month Patient education attention-control (AC) intervention includes 6 transplant educational materials, covering healthy post-transplant behavior, developed by the International Transplant Nurses Society. The RA calls Pps at 1, 2, 3, 4, 5 and 6 months to review the brochure information and answer any questions about it.
  Arms: Patient-education attention-control

SUMMARY:
With kidney transplant (KT) recipients as our exemplar population, our goal is to develop and test interventions that increase medication adherence (MA) in chronically ill adults. Among adult KT recipients, non-adherence to immunosuppressive medications (MNA) is the leading predictor of poor outcomes, including rejection, kidney loss, and death. An alarming one-third of KT patients experience MNA even though the problem is preventable. Adherence intervention studies have proven marginally effective for those with acute and chronic illnesses and ineffective for adult KT recipients. Using a randomized controlled trial design with an attention-control group, this R01 will test an innovative 6-month SystemCHANGE intervention to enhance immunosuppressive MA in adult non-adherent KT recipients. This intervention shows great promise for increasing MA with a large effect size of 1.4 in our pilot study. Grounded in the socio-ecological model, SystemCHANGE seeks to systematically improve MA behaviors by identifying and shaping routines, involving supportive others in routines, and using medication taking feedback through small patient-lead experiments to change and maintain behavior. The Medication Event Monitoring System cap, which contains microelectronics that record the date and time of the cap removal, will be used to measure MA. Persistence of the MA behavior change will be examined by evaluating the difference in MA between the two groups during the 6-month maintenance phase. Mediators and moderators of MA will be examined. Health outcomes will be compared and a cost-effectiveness analysis will be conducted.

DETAILED DESCRIPTION:
SPECIFIC AIMS For adult kidney transplant (KT) patients, the leading predictor of rejection, kidney loss, death and their attendant costs is immunosuppressive medications nonadherence (MNA). An alarming one-third of KT recipients experience this preventable problem. According to meta-analysis, predictors of MNA are nonwhite ethnicity, poorer social support and poorer perceived health. Patients' most frequent barrier to adhering to immunosuppressive medication is forgetting. 9 Even minor deviations from adherence have shown negative effects, though the precise extent of poor outcomes stemming from nonadherence is not clear. Traditionally, intervention studies aimed at boosting adherence target cognition (knowledge, attitudes, beliefs) and behavioral skills. However, these have proven marginally effective for individuals with acute and chronic illnesses and ineffective for adult KT recipients. In a sample of KT recipients, we propose to test the innovative and successful SystemCHANGE intervention, which is grounded in the socio-ecological model. This approach is a paradigm shift in behavioral interventions because it seeks to redesign the system of the interpersonal environment and daily routines linked to health behavior, rather than to alter individuals' efforts to change their behavior. Using a four-pronged, patient-centered approach, we will (1) assess individual systems (including important others who shape medication taking), how they influence medication taking and their proposals for improving medication adherence, (2) implement the proposed individual systems solutions for improving adherence, (3) track adherence data, and (4) evaluate adherence data through small experiments. In our pilot study, this intervention yielded a large effect size of 1.4.

This study's innovation lies in its use of a socio-ecological model known as SystemCHANGE, which differs greatly from previous cognitive and behavioral skills-focused interventions for improving medication adherence. This will be the first rigorous evaluation of SystemCHANGE with a diverse sample of KT recipients and long-term follow up. This study presents a unique opportunity to evaluate moderators and mediators of adherence and has potential, based upon pilot work, to have immediate "dose" impact. As such, it could hold great promise as an intervention that translates very well into practice settings. Our 6-month SystemCHANGE intervention (also referred to as "intervention") seeks to enhance adherence to immunosuppressive medication among adult KT recipients who are non-adherent. The study is a randomized controlled trial with an attention-control intervention (also referred to as "control") to determine persistence of medication adherence behavior change and differences in adherence between the two groups during the 6-month maintenance phase.

Primary Aim (PA):

PA: To determine whether the intervention is more effective than control in increasing medication adherence in adult KT recipients at the completion of the intervention and maintenance phases.

Hypothesis: Adult KT recipients participating in the intervention will have higher immunosuppressive adherence rates than those participating in the control at the completion of intervention and maintenance phases.

Secondary Aim (Sec):

SA: To examine the patterns of medication adherence in adult KT recipients in both groups.

Research question (RQ): When does the intervention become effective (e.g., what "dose" is needed)? RQ: What is the pattern of decay in adherence over time in both groups?

Exploratory Aims (EA):

EA1: To determine whether the intervention is more effective than the control in decreasing poor health outcomes (e.g. increasing creatinine/BUN, infection, acute/chronic rejection, graft loss, death, hospitalizations, length of hospital stay, and healthcare appointments).

Hypothesis: At one year, there will be differential levels of poor outcomes, with the intervention demonstrating lower levels of poor outcomes than the control.

EA2: To evaluate the role of potential mediators and moderators of medication adherence and health outcomes in adult KT recipients in the intervention and those in the control.

Hypothesis: Incorporating potential mediators and moderators of the intervention (e.g., nonwhite ethnicity, perceived social support, perceived health status, personal systems behavior) will increase the medication adherence variance explained by the intervention.

EA3: To determine if the intervention is cost-effective. Hypothesis: The cost-effectiveness ratio for the intervention will be less than for the control.

Each year, 35.6 KT recipients per 100 are non-adherent with their medications, which is the primary cause of post-transplant morbidity. Thus, the need for effective interventions is compelling: Decreasing transplant complications from MNA will reduce costs and make additional kidneys available to those waiting for transplants by reducing the number of KT recipients who must rejoin the organ list. This project builds on our research team's previous adherence work, including a SystemCHANGE intervention pilot study that addresses Healthy People 2020 initiatives of reducing chronic kidney disease complications, disability, death, and costs by optimizing transplant medication adherence and increasing the number of patients who receive a transplant.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 years or older,
2. prescribed at least 1 immunosuppressive medication taken twice a day,
3. functioning KT (not on dialysis),
4. has received a kidney-only transplant,
5. agreement from the transplant physician and nephrologist that individual is able to participate in the study,
6. able to speak, hear, and understand English as determined by the ability to participate and comprehend conversation about potential inclusion in the study,
7. able to open a MEMS cap as assessed by the Research Assistant (RA) asking if there is any problem with opening pill bottle caps,
8. able to administer immunosuppressive medications to self,
9. has a telephone or has access to a telephone,
10. has no cognitive impairment as determined by a score of 4 or greater on the 6-item Telephone Mental Status Screen Derived from the Mini-Mental Status Exam,
11. has no other diagnoses that may shorten life span, such as metastatic cancer,
12. is not currently hospitalized,
13. receives post-transplant care by the Missouri or Tennessee transplant programs.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2014-06; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Medication Adherence Change from Baseline to 6 Months | 6 months
  Medication adherence score of .85 or greater
Medication Adherence Change from 6 Months to 12 Months | 12 months
  Medication adherence score of .85 or greater
Medication Adherence Change from Baseline to 12 Months | 12
  Medication adherence score of .85 or greater

SECONDARY OUTCOMES:
Creatinine | 12 months
  Creatinine blood level
Infection | 12 months
  Blood, sputum, and/or urine culture positive for an abnormal organism
Acute rejection | 12 months
  Biposy proven
Chronic rejection | 12 months
  Biopsy proven
BUN | 12 months
  BUN blood level
Kidney graph loss | 12 months
  3-day dose of intravenous prednisone
Death | 12 months
  Death documented by transplant team
Cost effectiveness | 12 months
  Resource use costs of both Interventions

CONTACTS AND LOCATIONS:
Locations (1):
- University of Missouri-Kansas City, Kansas City, Missouri, United States

REFERENCES:
- [Derived] Mellon L, Doyle F, Hickey A, Ward KD, de Freitas DG, McCormick PA, O'Connell O, Conlon P. Interventions for increasing immunosuppressant medication adherence in solid organ transplant recipients. Cochrane Database Syst Rev. 2022 Sep 12;9(9):CD012854. doi: 10.1002/14651858.CD012854.pub2. PMID 36094829
- [Derived] Russell CL, Hathaway D, Remy LM, Aholt D, Clark D, Miller C, Ashbaugh C, Wakefield M, Ye S, Staggs VS, Ellis RJ, Goggin K. Improving medication adherence and outcomes in adult kidney transplant patients using a personal systems approach: SystemCHANGE results of the MAGIC randomized clinical trial. Am J Transplant. 2020 Jan;20(1):125-136. doi: 10.1111/ajt.15528. Epub 2019 Aug 20. PMID 31291507
- [Derived] Russell CL, Moore S, Hathaway D, Cheng AL, Chen G, Goggin K. MAGIC Study: Aims, Design and Methods using SystemCHANGE to Improve Immunosuppressive Medication Adherence in Adult Kidney Transplant Recipients. BMC Nephrol. 2016 Jul 16;17(1):84. doi: 10.1186/s12882-016-0285-8. PMID 27421884